CLINICAL TRIAL: NCT00421291
Title: Effect of Information on Service Delivery in Rural India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: World Bank (Other); Sahbhagi Shikshan Kendra (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: NA_00001063
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Delivery of Services to Rural Populations in India
MeSH Terms: interventions — Educational Status

INTERVENTIONS:
Behavioral: Education

SUMMARY:
A lack of public awareness about entitled health and social services may contribute to poor delivery of services in developing countries. We sought to determine the impact of educating villagers about entitled services.

DETAILED DESCRIPTION:
105 gram panchayats (village clusters) were randomized to receive information about their guaranteed health, education, and village governance rights. We then selected households within each treatment and control village to assess whether the information had made an impact.

ELIGIBILITY:
Inclusion Criteria:

* Gram panchayats in Uttar Pradesh

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-04; Study Completion 2005-10

PRIMARY OUTCOMES:
visits by nurse midwife
prenatal exams, tetanus vaccinations, & iron tablets received by pregnant women
infant vaccinations
educational scholarships and fees for children
occurrence of village council meetings
development work in villages

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Pandey, PhD, Principal Investigator — World Bank
Locations (1):
- No facility, this is a community based trial, Multiple Villages, Uttar Pradesh, India

REFERENCES:
- [Derived] Pandey P, Sehgal AR, Riboud M, Levine D, Goyal M. Informing resource-poor populations and the delivery of entitled health and social services in rural India: a cluster randomized controlled trial. JAMA. 2007 Oct 24;298(16):1867-75. doi: 10.1001/jama.298.16.1867. PMID 17954538